CLINICAL TRIAL: NCT01491113
Title: Single-Dose Pharmacokinetics of Orally Administered Levetiracetam (LEV) in Japanese Subjects With Normal Renal Function and Various Degrees of Renal Impairment Using a Dosing Regimen Adjusted to Renal Function (250 mg or 500 mg)
Brief Title: Pharmacokinetic (PK) Study in Japanese Non-epileptic Renal Impaired Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: N01373
Record Dates: First submitted 2011-12-09; First posted 2011-12-13 (Estimated); Results first posted 2014-01-10 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Healthy Subjects; Renal Impairments
Keywords: Levetiracetam; Oral administration; Japanese; Non-epileptic; Healthy; Renal impaired subjects
MeSH Terms: interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group A: Normal renal function (Experimental): Subjects who have normal renal function (CLcr >80 mL/min/1.73 m^2). Subjects will be orally administered Levetiracetam (LEV) 500 mg once. After LEV administration, safety assessments and blood and urine samplings will be taken through to Day 4 during the Treatment Period, and safety follow-up assessments will be performed on Day 8 according to the schedule of study assessments.
  * Blood samples for Pharmacokinetics (PK): Predose (Baseline), and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours postdose
  * Urine samples for PK: 0 - 6, 6 - 12, 12 - 24, 24 - 48, 48 - 72 hours postdose
  Interventions: Drug: Levetiracetam 500 mg
- Group B: Mild renal impairment (Experimental): Patients who have mild renal impairment (50<CLcr <80 mL/min/1.73 m^2). Subjects will be orally administered (Levetiracetam) LEV 500 mg once. After LEV administration, safety assessments and blood and urine samplings will be conducted through Day 5 during the Treatment Period, and safety follow-up assessments will be performed on Day 8 according to the schedule of study assessments.
  * Blood samples for Pharmacokinetics (PK): Predose (Baseline), and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96 hours postdose
  * Urine samples for PK: 0 - 6, 6 - 12, 12 - 24, 24 - 48, 48 - 72, 72 - 96 hours postdose
  Interventions: Drug: Levetiracetam 500 mg
- Group C: Moderate renal impairment (Experimental): Patients who have moderate renal impairment (30<CLcr < 50 mL/min/1.73 m^2). Subjects will be orally administered Levetiracetam (LEV) 250 mg once. After LEV administration, safety assessments and blood and urine samplings will be conducted through Day 6 during the Treatment Period, and safety follow-up assessments will be performed on Day 8 according to the schedule of study assessments.
  * Blood samples for Pharmacokinetics (PK): Predose (Baseline), and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours postdose
  * Urine samples for PK: 0 - 6, 6 - 12, 12 - 24, 24 - 48, 48 - 72, 72 - 96, 96 -120 hours postdose
  Interventions: Drug: Levetiracetam 250 mg
- Group D: Severe renal impairment (Experimental): Patients who have severe renal impairment (CLcr <30 mL/min/1.73 m^2). Subjects will be orally administered Levetiracetam (LEV) 250 mg once. After LEV administration, safety assessments and blood and urine samplings will be conducted through Day 7 during the Treatment Period, and safety follow-up assessments will be performed on Day 8 according to the schedule of study assessments.
  * Blood samples for Pharmacokinetics (PK): Predose (Baseline), and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144 hours postdose
  * Urine samples for PK: 0 - 6, 6 - 12, 12 - 24, 24 - 48, 48 - 72, 72 - 96, 96 -120, 120 - 144 hours postdose
  Interventions: Drug: Levetiracetam 250 mg
- Group E: End-stage renal disease (Experimental): Group E will receive Levetiracetam (LEV) 500 mg on Day 1, 44 hours (h) before the first hemodialysis. As a supplementary dose LEV 250 mg will be administered 1 h after the end of the first hemodialysis on Day 3.
  The 4-h Hemodialysis are scheduled as follows:
  1. Dialysis: 44 h to 48 h after the first dose (Day 3)
  2. Dialysis: 92 h to 96 h after the first dose (Day 5)
  3. Dialysis: 140 h after the first dose (Day 7)
  Safety assessments and blood samplings will be conducted until Day 7. Safety follow-up assessments will be performed on Day 10.
  Blood samples for Pharmacokinetics (PK): Predose (Baseline), and 0.5, 1, 2, 4, 6, 8, 12, 24, 30, 44*, 44.25*, 44.5*, 45*, 46*, 47*, 48*, 49, 49.5, 50, 51, 53, 55, 57, 61, 73, 92, 96, 120, 140 hours post first dosing.
  49 h-sample should be taken before the additional dose. The 44 h, 92 h, and 140 h sample should be taken before the start of the hemodialysis.
  *Inflow blood, outflow blood, and dialysate fluid will be collected.
  Interventions: Drug: Levetiracetam 250 mg; Drug: Levetiracetam 500 mg

INTERVENTIONS:
Drug: Levetiracetam 250 mg — Tablet containing Levetiracetam 250 mg
  Other Names: E-Keppra
  Arms: Group C: Moderate renal impairment; Group D: Severe renal impairment; Group E: End-stage renal disease
Drug: Levetiracetam 500 mg — Tablet containing Levetiracetam 500 mg
  Other Names: E-Keppra
  Arms: Group A: Normal renal function; Group B: Mild renal impairment; Group E: End-stage renal disease

SUMMARY:
This is a human pharmacology, single-dose study to investigate the pharmacokinetics of orally administered Levetiracetam (LEV) in Japanese subjects with normal renal function and in Japanese subjects with various degrees of impaired renal function.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the plasma and urine PK of Levetiracetam (ucb L059) and its metabolite (ucb L057) after a single dose of LEV 250 mg or LEV 500 mg in Japanese subjects with normal renal function and in Japanese subjects with various degrees of renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with normal renal function
* Subject is Japanese
* Subjects with creatinine clearance within 1 of 3 Groups (CLcr[mL/min/1.73 cm^2]: Group B: 50 - <80, Group C: 30 - <50, Group D: <30), or for Group E, subjects with end-stage renal failure undergoing hemodialysis

Exclusion Criteria:

* Subjects has taken any drug treatment, disease or injury to influence Levetiracetam PK except for renal impairments

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (2):
- Japan (2):
  - 1, Fukuoka
  - 2, Ibaraki

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Participant Flow refers to the Safety Set population which includes all patients that received at least one dose of study medication.
Pre-assignment Details: About 30 (28 to 30) subjects were planned to be enrolled for 5 groups (A to E) according to their renal function based on the value of creatinine clearance (CLCr).
Groups:
- Group A: Normal Renal Function: Subjects with normal renal function (CLcr >80 mL/min/1.73 m^2). Subjects were orally administered Levetiracetam (LEV) 500 mg once. After LEV administration, safety assessments and blood and urine samplings were taken through to Day 4 during the Treatment Period, and safety follow-up assessments were performed on Day 8 according to the schedule of study assessments.
  * Blood samples for Pharmacokinetic (PK) analyses: Predose (Baseline), and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72 hours postdose
  * Urine samples for PK analyses: 0 - 6, 6 - 12, 12 - 24, 24 - 48, 48 - 72 hours postdose
- Group B: Mild Renal Impairment: Patients with mild renal impairment (50<CLcr <80 mL/min/1.73 m^2). Subjects were orally administered (Levetiracetam) LEV 500 mg once. After LEV administration, safety assessments and blood and urine samplings were conducted through Day 5 during the Treatment Period, and safety follow-up assessments were performed on Day 8 according to the schedule of study assessments.
  * Blood samples for Pharmacokinetic (PK) analyses: Predose (Baseline), and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96 hours postdose
  * Urine samples for PK analyses: 0 - 6, 6 - 12, 12 - 24, 24 - 48, 48 - 72, 72 - 96 hours postdose
- Group C: Moderate Renal Impairment: Patients with moderate renal impairment (30<CLcr < 50 mL/min/1.73 m^2). Subjects were orally administered Levetiracetam (LEV) 250 mg once. After LEV administration, safety assessments and blood and urine samplings were conducted through Day 6 during the Treatment Period, and safety follow-up assessments were performed on Day 8 according to the schedule of study assessments.
  * Blood samples for Pharmacokinetic (PK) analyses: Predose (Baseline), and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours postdose
  * Urine samples for PK analyses: 0 - 6, 6 - 12, 12 - 24, 24 - 48, 48 - 72, 72 - 96, 96 -120 hours postdose
- Group D: Severe Renal Impairment: Patients with severe renal impairment (CLcr <30 mL/min/1.73 m^2). Subjects were orally administered Levetiracetam (LEV) 250 mg once. After LEV administration, safety assessments and blood and urine samplings were conducted through Day 7 during the Treatment Period, and safety follow-up assessments were performed on Day 8 according to the schedule of study assessments.
  * Blood samples for Pharmacokinetic (PK) analyses: Predose (Baseline), and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144 hours postdose
  * Urine samples for PK analyses: 0 - 6, 6 - 12, 12 - 24, 24 - 48, 48 - 72, 72 - 96, 96 -120, 120 - 144 hours postdose
- Group E: End-stage Renal Disease: Group E received Levetiracetam (LEV) 500 mg orally on Day 1, 44 hours (h) before the first hemodialysis. As a supplementary dose LEV 250 mg was administered 1 h after the end of the first hemodialysis on Day 3.
  The 4-h Hemodialysis was scheduled as follows:
  1. Dialysis: 44 h to 48 h after the first dose (Day 3)
  2. Dialysis: 92 h to 96 h after the first dose (Day 5)
  3. Dialysis: 140 h after the first dose (Day 7)
  Safety assessments and blood samplings were conducted until Day 7. Safety follow-up assessments were performed on Day 10.
  Blood samples for Pharmacokinetics (PK): Predose (Baseline), and 0.5, 1, 2, 4, 6, 8, 12, 24, 30, 44*, 44.25*, 44.5*, 45*, 46*, 47*, 48*, 49, 49.5, 50, 51, 53, 55, 57, 61, 73, 92, 96, 120, 140 hours post first dosing.
  49 h-sample was taken before the additional dose. The 44 h, 92 h, and 140 h samples were taken before the start of the hemodialysis.
  *Inflow blood, outflow blood, and dialysate fluid were collected.
Period: Overall Study
Arm/Group | Group A: Normal Renal Function | Group B: Mild Renal Impairment | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment | Group E: End-stage Renal Disease
Started | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population refers to the Pharmacokinetic Per Protocol Set (PK-PPS) which consists of all subjects included in the Safety Set (SS), who also had a sufficient number of bioanalytical assessments (plasma or urine) to calculate reliable estimates for the PK parameters.
Groups:
- Group B: Mild Renal Impairment: Patients with mild renal impairment (50<CLcr <80 mL/min/1.73 m^2). Subjects were orally administered (Levetiracetam) LEV 500 mg once. After LEV administration, safety assessments and blood and urine samplings were conducted through Day 5 during the Treatment Period, and safety follow-up assessments were performed on Day 8 according to the schedule of study assessments.
  * Blood samples for Pharmacokinetics (PK) analyses: Predose (Baseline), and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96 hours postdose
  * Urine samples for PK analyses: 0 - 6, 6 - 12, 12 - 24, 24 - 48, 48 - 72, 72 - 96 hours postdose
- Group E: End-stage Renal Disease: Group E received Levetiracetam (LEV) 500 mg orally on Day 1, 44 hours (h) before the first hemodialysis. As a supplementary dose LEV 250 mg was administered 1 h after the end of the first hemodialysis on Day 3.
  The 4-h Hemodialysis was scheduled as follows:
  1. Dialysis: 44 h to 48 h after the first dose (Day 3)
  2. Dialysis: 92 h to 96 h after the first dose (Day 5)
  3. Dialysis: 140 h after the first dose (Day 7)
  Safety assessments and blood samplings were conducted until Day 7. Safety follow-up assessments were performed on Day 10.
  Blood samples for Pharmacokinetic (PK) analyses: Predose (Baseline), and 0.5, 1, 2, 4, 6, 8, 12, 24, 30, 44*, 44.25*, 44.5*, 45*, 46*, 47*, 48*, 49, 49.5, 50, 51, 53, 55, 57, 61, 73, 92, 96, 120, 140 hours post first dosing.
  49 h-sample was taken before the additional dose. The 44 h, 92 h, and 140 h samples were taken before the start of the hemodialysis.
  *Inflow blood, outflow blood, and dialysate fluid were collected.
- Total: Total of all reporting groups
Arm/Group | Group A: Normal Renal Function | Group B: Mild Renal Impairment | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment | Group E: End-stage Renal Disease | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (2.6) | 67.5 (5.0) | 69.3 (6.1) | 55.8 (17.1) | 68.8 (7.9) | 64.6 (10.0)
Age, Customized [Number; unit: participants]
  20 - <65 years | 5 | 3 | 1 | 4 | 2 | 15
  >=65 years | 1 | 3 | 5 | 2 | 4 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 0 | 0 | 1
  Male | 5 | 6 | 6 | 6 | 6 | 29
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 6 | 6 | 6 | 6 | 6 | 30
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 6 | 6 | 6 | 6 | 6 | 30
Weight [Mean (Standard Deviation); unit: kilogram] | 60.95 (10.97) | 74.28 (4.14) | 63.07 (12.49) | 58.70 (6.10) | 62.20 (5.41) | 63.84 (9.62)
Height [Mean (Standard Deviation); unit: centimeters] | 161.73 (9.05) | 165.65 (3.11) | 163.72 (5.64) | 164.50 (6.34) | 162.38 (3.41) | 163.60 (5.68)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ucb L059 (LEV) for Groups A to D
Description: Cmax refers to the maximum observed concentration of L059 (Levetiracetam).
  Group A: Baseline to 72 hours; Group B: Baseline to 96 hours; Group C: Baseline to 120 hours; Group D: Baseline to 144 hours
Time Frame: From Baseline up to 144 hours post first dose
Population: The Analysis Population refers to the Pharmacokinetic Per Protocol Set which consists of all subjects included in the Safety Set, who also have a sufficient number of bioanalytical assessments (plasma or urine) to calculate reliable estimates for the Pharmacokinetic parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Group A: Normal Renal Function | Group B: Mild Renal Impairment | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
µg/mL | 21.9357 (31.2) | 15.5334 (25.3) | 10.7767 (24.3) | 9.1754 (30.4)

2. Primary Outcome: Area Under the Concentration-time Curve (AUC(0-t)) of Ucb L059 (LEV) From Baseline to the Last Quantifiable Concentration for Groups A to D
Description: AUC(0-t) refers to the area under the plasma concentration versus time curve, which provides information on the exposure.
  Group A: Baseline to 72 hours; Group B: Baseline to 96 hours; Group C: Baseline to 120 hours; Group D: Baseline to 144 hours
Time Frame: From Baseline up to 144 hours post first dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | Group A: Normal Renal Function | Group B: Mild Renal Impairment | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
h*µg/mL | 165.9996 (16.5) | 247.6430 (16.9) | 169.3392 (16.5) | 212.1193 (19.1)

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ucb L057 for Groups A to D
Description: Cmax refers to the maximum observed concentration of ucb L057.
  Group A: Baseline to 72 hours; Group B: Baseline to 96 hours; Group C: Baseline to 120 hours; Group D: Baseline to 144 hours
Time Frame: From Baseline up to 144 hours post first dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Group A: Normal Renal Function | Group B: Mild Renal Impairment | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
µg/mL | 0.3620 (9.4) | 0.7503 (25.8) | 0.5674 (26.0) | 1.0640 (29.3)

4. Primary Outcome: Area Under the Concentration-time Curve (AUC(0-t)) of Ucb L057 From Baseline to the Last Quantifiable Concentration for Groups A to D
Description: as for outcome 2
Time Frame: From Baseline up to 144 hours post first dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | Group A: Normal Renal Function | Group B: Mild Renal Impairment | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
h*µg/mL | 5.8607 (9.7) | 22.5573 (45.9) | 18.6675 (53.4) | 57.7773 (57.3)

5. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ucb L059 (LEV) for Group E During First Period
Description: Cmax refers to the maximum observed concentration of ucb L059 (Levetiracetam).
Time Frame: From Baseline to 44 hours post first dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Group E: End-stage Renal Disease
Number analyzed (Participants) | 6
µg/mL | 18.6810 (8.1)

6. Primary Outcome: Area Under the Concentration-time Curve (AUC(0-t)) of Ucb L059 (LEV) From Baseline to 44 Hours for Group E
Description: AUC(0-t) refers to the area under the plasma concentration versus time curve, which provides information on the exposure.
Time Frame: From Baseline to 44 hours post first dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | Group E: End-stage Renal Disease
Number analyzed (Participants) | 6
h*µg/mL | 462.4883 (10.5)

7. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ucb L057 for Group E During First Period
Description: Cmax refers to the maximum observed concentration of ucb L057.
Time Frame: From Baseline to 44 hours post first dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- Group E: End-stage Renal Disease: Group E received Levetiracetam (LEV) 500 mg orally on Day 1, 44 hours (h) before the first hemodialysis. As a supplementary dose LEV 250 mg was administered 1 h after the end of the first hemodialysis on Day 3.
  The 4-h Hemodialysis was scheduled as follows:
  1. Dialysis: 44 h to 48 h after the first dose (Day 3)
  2. Dialysis: 92 h to 96 h after the first dose (Day 5)
  3. Dialysis: 140 h after the first dose (Day 7)
  Safety assessments and blood samplings were conducted until Day 7. Safety follow-up assessments were performed on Day 10.
  Blood samples for Pharmacokinetics (PK) analyses: Predose (Baseline), and 0.5, 1, 2, 4, 6, 8, 12, 24, 30, 44*, 44.25*, 44.5*, 45*, 46*, 47*, 48*, 49, 49.5, 50, 51, 53, 55, 57, 61, 73, 92, 96, 120, 140 hours post first dosing.
  49 h-sample was taken before the additional dose. The 44 h, 92 h, and 140 h samples were taken before the start of the hemodialysis.
  *Inflow blood, outflow blood, and dialysate fluid were collected.
Arm/Group | Group E: End-stage Renal Disease
Number analyzed (Participants) | 6
µg/mL | 8.8435 (7.0)

8. Primary Outcome: Area Under the Concentration-time Curve (AUC(0-t)) of Ucb L057 From Baseline to 44 Hours for Group E
Description: as for outcome 6
Time Frame: From Baseline to 44 hours post first dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | Group E: End-stage Renal Disease
Number analyzed (Participants) | 6
h*µg/mL | 230.4393 (7.8)

9. Secondary Outcome: Total Amount Excreted in Urine (Ae) of Ucb L059 (LEV) for Groups A to D
Description: Ae refers to the total amount of ucb L059 (Levetiracetam) excreted in urine.
  Group A: Baseline to 72 hours; Group B: Baseline to 96 hours; Group C: Baseline to 120 hours; Group D: Baseline to 144 hours
Time Frame: From Baseline up to 144 hours post first dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Group A: Normal Renal Function | Group B: Mild Renal Impairment | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment
Number analyzed (Participants) | 4 | 6 | 6 | 6
mg | 304.7321 (30.3) | 247.6562 (12.5) | 98.7182 (11.9) | 74.3761 (34.4)

10. Secondary Outcome: Fraction of Dose Excreted in Urine (fe) of Ucb L059 (LEV) for Groups A to D
Description: fe refers to the fraction of dose excreted in urine of L059 (Levetiracetam).
  Group A: Baseline to 72 hours; Group B: Baseline to 96 hours; Group C: Baseline to 120 hours; Group D: Baseline to 144 hours
Time Frame: From Baseline up to 144 hours post first dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of Dose Administered
Arm/Group | Group A: Normal Renal Function | Group B: Mild Renal Impairment | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment
Number analyzed (Participants) | 4 | 6 | 6 | 6
Percentage of Dose Administered | 60.9464 (30.3) | 49.5312 (12.5) | 39.4873 (11.9) | 29.7504 (34.4)

11. Secondary Outcome: Renal Clearance (CLR) of Ucb L059 (LEV) for Groups A to D
Description: Renal clearance describes the removal of drug from a volume of plasma in a given unit of time by the kidneys.
  Group A: Baseline to 72 hours; Group B: Baseline to 96 hours; Group C: Baseline to 120 hours; Group D: Baseline to 144 hours
Time Frame: From Baseline up to 144 hours post first dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Group A: Normal Renal Function | Group B: Mild Renal Impairment | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment
Number analyzed (Participants) | 4 | 6 | 6 | 6
L/h | 1.8622 (27.4) | 0.9820 (22.1) | 0.5671 (17.6) | 0.3417 (49.3)

12. Secondary Outcome: Apparent Total Body Clearance (CL/F) of Ucb L059 (LEV) for Groups A to D
Description: Clearance (expressed as volume/time) describes the removal of drug from a volume of plasma in a given unit of time (drug loss from the body). It indicates the volume of plasma (or blood) from which the drug is completely removed, or cleared, in a given time period.
  Group A: Baseline to 72 hours; Group B: Baseline to 96 hours; Group C: Baseline to 120 hours; Group D: Baseline to 144 hours
Time Frame: From Baseline up to 144 hours post first dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Group A: Normal Renal Function | Group B: Mild Renal Impairment | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
L/h | 2.9359 (14.8) | 1.9826 (16.0) | 1.4362 (15.3) | 1.1484 (19.1)

13. Secondary Outcome: Nonrenal Clearance (CLNR) of Ucb L059 (LEV) for Groups A to D
Description: The Non-Renal Clearance (CLNR) describes the removal of drug by organs other than the kidneys.
  Group A: Baseline to 72 hours; Group B: Baseline to 96 hours; Group C: Baseline to 120 hours; Group D: Baseline to 144 hours
Time Frame: From Baseline up to 144 hours post first dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Group A: Normal Renal Function | Group B: Mild Renal Impairment | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment
Number analyzed (Participants) | 4 | 6 | 6 | 6
L/h | 1.0712 (50.6) | 0.9873 (17.4) | 0.8636 (18.4) | 0.7848 (17.9)

14. Secondary Outcome: Total Amount Excreted in Urine (Ae) of Ucb L057 for Groups A to D
Description: Ae refers to the total amount of ucb L057 excreted in urine.
  Group A: Baseline to 72 hours; Group B: Baseline to 96 hours; Group C: Baseline to 120 hours; Group D: Baseline to 144 hours
Time Frame: From Baseline up to 144 hours post first dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Group A: Normal Renal Function | Group B: Mild Renal Impairment | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment
Number analyzed (Participants) | 4 | 6 | 6 | 6
mg | 83.5936 (16.9) | 169.3395 (19.0) | 93.1346 (14.0) | 100.7489 (17.8)

15. Secondary Outcome: Renal Clearance (CLR) of Ucb L057 for Groups A to D
Description: as for outcome 11
Time Frame: From Baseline up to 144 hours post first dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Group A: Normal Renal Function | Group B: Mild Renal Impairment | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment
Number analyzed (Participants) | 4 | 6 | 6 | 6
L/h | 14.6937 (18.3) | 6.8015 (32.6) | 4.6828 (45.6) | 1.6475 (42.0)

16. Secondary Outcome: Apparent Total Body Clearance (CL/F) of Ucb L059 (LEV) for Group E During First Period
Description: Clearance (expressed as volume/time) describes the removal of drug from a volume of plasma in a given unit of time (drug loss from the body). It indicates the volume of plasma (or blood) from which the drug is completely removed, or cleared, in a given time period.
  Geometric mean and Coefficient of Variation (CV) was not calculated since the extrapolated part of the AUC was greater than 20 %.
Time Frame: From Baseline to 44 hours post first dose
Population: as for outcome 1
Measure: Median (Full Range); unit: L/h
Arm/Group | Group E: End-stage Renal Disease
Number analyzed (Participants) | 6
L/h | 0.629 [0.500 to 0.801]

17. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Ucb L059 (LEV) for Groups A to D
Description: tmax refers to the time to reach maximum plasma concentration of ucb L059 (Levetiracetam).
  Group A: Baseline to 72 hours; Group B: Baseline to 96 hours; Group C: Baseline to 120 hours; Group D: Baseline to 144 hours
Time Frame: From Baseline up to 144 hours post first dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Group A: Normal Renal Function | Group B: Mild Renal Impairment | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours | 0.500 [0.500 to 2.000] | 1.000 [0.500 to 2.000] | 0.500 [0.500 to 1.000] | 0.500 [0.500 to 1.000]

18. Secondary Outcome: Area Under the Concentration-time Curve (AUC) of Ucb L059 (LEV) From Baseline to Infinite for Groups A to D
Description: as for outcome 2
Time Frame: From Baseline up to 144 hours post first dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | Group A: Normal Renal Function | Group B: Mild Renal Impairment | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
h*µg/mL | 170.3045 (14.8) | 252.1923 (16.0) | 174.0764 (15.3) | 217.6854 (19.1)

19. Secondary Outcome: Terminal Half-life (t1/2) of Ucb L059 (LEV) for Groups A to D
Description: Terminal half-life refers to the time it takes for the concentrations to decrease by half.
  Group A: Baseline to 72 hours; Group B: Baseline to 96 hours; Group C: Baseline to 120 hours; Group D: Baseline to 144 hours
Time Frame: From Baseline up to 144 hours post first dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group A: Normal Renal Function | Group B: Mild Renal Impairment | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours | 7.6164 (6.9) | 12.6214 (11.3) | 15.5033 (17.5) | 19.7320 (26.5)

20. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Ucb L057 for Groups A to D
Description: tmax refers to the time to reach maximum plasma concentration (tmax).
  Group A: Baseline to 72 hours; Group B: Baseline to 96 hours; Group C: Baseline to 120 hours; Group D: Baseline to 144 hours
Time Frame: From Baseline up to 144 hours post first dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Group A: Normal Renal Function | Group B: Mild Renal Impairment | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours | 5.000 [2.000 to 8.000] | 8.000 [6.000 to 12.000] | 12.000 [8.000 to 12.000] | 24.000 [12.000 to 24.000]

21. Secondary Outcome: Area Under the Concentration-time Curve (AUC) of Ucb L057 From Baseline to Infinite for Groups A to D
Description: AUC(0-t) refers to the area under the plasma concentration versus time curve, which provides information on the exposure.
  Geometric mean and CV was not calculated since the extrapolated part of the AUC was greater than 20 %.
  Group A: Baseline to 72 hours; Group B: Baseline to 96 hours; Group C: Baseline to 120 hours; Group D: Baseline to 144 hours
Time Frame: From Baseline up to 144 hours post first dose
Population: as for outcome 1
Measure: Median (Full Range); unit: h*µg/mL
Arm/Group | Group A: Normal Renal Function | Group B: Mild Renal Impairment | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment
Number analyzed (Participants) | 5 | 4 | 4 | 4
h*µg/mL | 8.176 (0) [7.432 to 11.085] | 32.401 [28.910 to 38.917] | 27.441 [16.472 to 41.184] | 63.126 [48.016 to 171.348]

22. Secondary Outcome: Terminal Half-life (t1/2) of Ucb L057 for Groups A to D
Description: as for outcome 19
Time Frame: From Baseline up to 144 hours post first dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Group A: Normal Renal Function | Group B: Mild Renal Impairment | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment
Number analyzed (Participants) | 5 | 4 | 4 | 4
hours | 12.351 [11.348 to 15.310] | 19.030 [17.331 to 19.903] | 20.303 [19.681 to 23.569] | 26.769 [17.249 to 33.348]

23. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Ucb L059 (Levetiracetam) for Group E During First Period
Description: tmax refers to the time to reach the maximum plasma concentration of ucb L059 (Levetiracetam).
Time Frame: From Baseline to 44 hours post first dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Group E: End-stage Renal Disease
Number analyzed (Participants) | 6
hours | 0.720 [0.430 to 0.980]

24. Secondary Outcome: Area Under the Concentration-time Curve (AUC) of Ucb L059 (LEV) From Baseline to Infinite for Group E
Description: AUC(0-t) refers to the area under the plasma concentration versus time curve, which provides information on the exposure.
  Geometric mean and CV was not calculated since the extrapolated part of the AUC was greater than 20 %.
Time Frame: From Baseline to 140 hours post first dose
Population: as for outcome 1
Measure: Median (Full Range); unit: h*µg/mL
Arm/Group | Group E: End-stage Renal Disease
Number analyzed (Participants) | 6
h*µg/mL | 794.588 (10.5) [624.521 to 999.853]

25. Secondary Outcome: Terminal Half-life (t1/2) of Ucb L059 (LEV) for Group E During First Period
Description: Terminal half-life refers to the time it takes for the concentrations to decrease by half.
  Geometric mean and CV was not calculated since the extrapolated part of the AUC was greater than 20 %.
Time Frame: From Baseline to 44 hours post first dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Group E: End-stage Renal Disease
Number analyzed (Participants) | 6
hours | 34.669 [29.227 to 38.648]

26. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Ucb L057 for Group E During First Period
Description: tmax refers to the time to reach maximum plasma concentration (tmax).
Time Frame: From Baseline to 44 hours post first dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Group E: End-stage Renal Disease
Number analyzed (Participants) | 6
hours | 44.020 [44.000 to 44.030]

27. Secondary Outcome: Hemodialysis Clearance (CLD) of Ucb L059 (LEV) During First Dialysis for Group E
Description: Calculated by the Arterio - Venous difference method and cumulative dialysate method.
Time Frame: From 44 hours to 48 hours post first dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Group E: End-stage Renal Disease
Number analyzed (Participants) | 6
mL/min | 113.9665 (8.5)

28. Secondary Outcome: Ultrafiltration Clearance (CLUF) of Ucb L059 (LEV) During First Dialysis for Group E
Description: Calculated by the Arterio - Venous difference method and cumulative dialysate method.
Time Frame: From 44 hours to 48 hours post first dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Group E: End-stage Renal Disease
Number analyzed (Participants) | 6
mL/min | 1.3271 (32.5)

29. Secondary Outcome: Hemodialysis Clearance (CLHD) of Ucb L059 (LEV) During First Dialysis for Group E
Description: Calculated according: CLHD=CLD+CLUF.
Time Frame: From 44 hours to 48 hours post first dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Groups:
- Group E: End-stage Renal Disease: Group E received Levetiracetam (LEV) 500 mg orally on Day 1, 44 hours (h) before the first hemodialysis. As a supplementary dose LEV 250 mg was administered 1 h after the end of the first hemodialysis on Day 3.
  The 4-h Hemodialysis was scheduled as follows:
  1. Dialysis: 44 h to 48 h after the first dose (Day 3)
  2. Dialysis: 92 h to 96 h after the first dose (Day 5)
  3. Dialysis: 140 h after the first dose (Day 7)
  Safety assessments and blood samplings were conducted until Day 7. Safety follow-up assessments were performed on Day 10.
  Blood samples for Pharmacokinetics (PK) analysis: Predose (Baseline), and 0.5, 1, 2, 4, 6, 8, 12, 24, 30, 44*, 44.25*, 44.5*, 45*, 46*, 47*, 48*, 49, 49.5, 50, 51, 53, 55, 57, 61, 73, 92, 96, 120, 140 hours post first dosing.
  49 h-sample was taken before the additional dose. The 44 h, 92 h, and 140 h samples were taken before the start of the hemodialysis.
  *Inflow blood, outflow blood, and dialysate fluid were collected.
Arm/Group | Group E: End-stage Renal Disease
Number analyzed (Participants) | 6
mL/min | 115.3702 (8.1)

ADVERSE EVENTS:
Time Frame: Treatment-Emergent Adverse Events were reported from Day 1 up to Day 8 (+2 days) for Group A to D and from Day 1 up to Day 10 (+2 days) for Group E.
Description: Treatment-Emergent Adverse Events (TEAEs) were reported. TEAEs are defined as those adverse events that either start or worsen in intensity on or after the date/time of first dose of study treatment.
Arm/Group | Group A: Normal Renal Function | Group B: Mild Renal Impairment | Group C: Moderate Renal Impairment | Group D: Severe Renal Impairment | Group E: End-stage Renal Disease
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 0/6 | 2/6 | 0/6 | 1/6 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Normal Renal Function (N=6) | Group B: Mild Renal Impairment (N=6) | Group C: Moderate Renal Impairment (N=6) | Group D: Severe Renal Impairment (N=6) | Group E: End-stage Renal Disease (N=6)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shunt malfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Normal Renal Function (N=6) | Group B: Mild Renal Impairment (N=6) | Group C: Moderate Renal Impairment (N=6) | Group D: Severe Renal Impairment (N=6) | Group E: End-stage Renal Disease (N=6)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days